CLINICAL TRIAL: NCT03598322
Title: The Volume Effect of Hydrodissection for Injection Therapies in Patients With Carpal Tunnel Syndrome - Evaluation Model by Shear Wave Ultrasound Elastography and Artificial Intelligence Imaging Analysis
Brief Title: The Volume Effect of Hydrodissection for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201711014RINA
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2017-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dextrose 1mL (Active Comparator): Dextrose injection, Dextrose 1mL, active comparator
  Interventions: Procedure: Dextrose 1mL injection
- Dextrose 2mL (Experimental): Dextrose injection, Dextrose 2mL
  Interventions: Procedure: Dextrose 2mL injection
- Dextrose 4mL (Experimental): 'Dextrose injection, Dextrose 4mL
  Interventions: Procedure: Dextrose 4mL injection

INTERVENTIONS:
Procedure: Dextrose 1mL injection — Dextrose 1mL injection and hydrodissection for CTS
  Arms: Dextrose 1mL
Procedure: Dextrose 2mL injection — Dextrose 2mL injection
  Arms: Dextrose 2mL
Procedure: Dextrose 4mL injection — Dextrose 4mL injection
  Arms: Dextrose 4mL

SUMMARY:
The investigators investigated the volume effect of hydrodissection for Injection therapies in patients with Carpal Tunnel Syndrome. The investigators evaluated participants by Shear Wave Ultrasound Elastography and Artificial Intelligence Imaging Analysis

DETAILED DESCRIPTION:
The investigators investigated the volume effect of hydrodissection for Injection therapies in patients with Carpal Tunnel Syndrome. The investigators evaluated participants by Shear Wave Ultrasound Elastography and Artificial Intelligence Imaging Analysis

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80
* Electrophysiological diagnosis of carpal tunnel syndrome
* At least one of the following two:

  1. Tenderness or numbness over median nerve innervated dermatome over 2 months
  2. Phalen test or Tinel sign or flick sign positive

Exclusion Criteria:

* History of wrist surgery
* Wrist trauma in recent two years
* Received wrist injection in recent three months
* History of brachial plexopathy, cervical radiculopathy or thoracic outlet syndrome
* History of DM, thyroid disorder or autoimmune disease
* Unable to cooperate with interview, examination or injection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Visual analog scale (VAS) | 1 week, 4 weeks, 12 weeks, 24 weeks
  Change of Visual analog scale (VAS), from Baseline

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire Score (BCTQ) | 1 week, 4 weeks, 12 weeks, 24 weeks
  Boston Carpal Tunnel Syndrome Questionnaire Score (BCTQ), 19 items with each item scale 1-5
QuickDASH | 1 week, 4 weeks, 12 weeks, 24 weeks
  QuickDASH (The Disabilities of the Arm, Shoulder and Hand Score(QuickDash)), 11 items with each item scale 1-5
MSK US finding | 1 week, 4 weeks, 12 weeks, 24 weeks
  Cross-sectional area of median nerve

CONTACTS AND LOCATIONS:
Overall Officials: Chueh Hung Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Physical Medicine & Rehabilitation , National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin MT, Liao CL, Hsiao MY, Hsueh HW, Chao CC, Wu CH. Volume Matters in Ultrasound-Guided Perineural Dextrose Injection for Carpal Tunnel Syndrome: A Randomized, Double-Blinded, Three-Arm Trial. Front Pharmacol. 2020 Dec 17;11:625830. doi: 10.3389/fphar.2020.625830. eCollection 2020. PMID 33391002